CLINICAL TRIAL: NCT01760239
Title: Electronic Health Record-Based Clinical Decision Support to Improve Blood Pressure Management in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-090; R01HL115082 (NIH)
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2017-06

CONDITIONS: Hypertension; Pre Hypertension; Obesity
Keywords: Adolescent Hypertension; Adolescent Pre Hypertension; Adolescent Pre Hypertension and Obesity
MeSH Terms: conditions — Hypertension; Prehypertension; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinical Decision Support (CDS) (Experimental): The Clinical Decision Support (CDS) tool will be activated when a BP is entered in the vital sign section of the EHR during any visit to a family practice or pediatric clinic (including both preventive care and sick visits, excluding prenatal and postpartum visits). The algorithm will be embedded in the EHR. In most cases, when a normal BP <90% and <120/80 mm Hg is entered, no alerts will be triggered. In some cases, clinical staff may receive up to two alerts, either to measure height or to repeat a first elevated BP reading. In cases with confirmed elevated BP measures, providers will receive a single CDS message summarizing that patient's current BP status and recommending specific clinical actions.
  Interventions: Behavioral: Clinical Decision Support (CDS)
- Control (No Intervention): Patients in this group will receive usual care from their clinic. The CDS tool will not be activated.

INTERVENTIONS:
Behavioral: Clinical Decision Support (CDS) — The Clinical Decision Support (CDS) tool will be activated when a BP is entered in the vital sign section of the EHR. The CDS tool includes six key features: (i) prompts regarding the need for height data to classify the BP by percentile (ii) prompts to repeat any BP that is ≥90% or ≥120/80 mm Hg (iii) classification of BPs by percentile, including classification of those in pre-HT, stage 1 HT and stage 2 HT range (iv) review of previous HT diagnoses and BPs in order to classify elevated BPs as incident (first or second elevated BP) or persistent (third or greater elevated BP) (v) tailored CDS based on HT category and previous diagnoses (vi) graphical representation of current and historical BP data by age and BP percentile.
  Arms: Clinical Decision Support (CDS)

SUMMARY:
The goal of this project is to improve detection and management of elevated blood pressure in adolescents. It (a) uses electronic health record (EHR) technology to deliver patient-specific clinical decision support (CDS) to providers at the point of care, (b) assesses the impact of this intervention on identification and clinical care of hypertension in adolescents, and (c) assesses the impact of the intervention on costs of care.

DETAILED DESCRIPTION:
Hypertension (HT) during adolescence tracks into adulthood, contributing to adult cardiovascular morbidity and mortality. National guidelines for the diagnosis and treatment of hypertension in children and adolescents were developed by the National High Blood Pressure Education Program (NHBPEP); their Fourth Report was published in 2004. Despite heightened awareness of hypertension in pediatric populations, most adolescents with elevated blood pressure remain clinically unrecognized. Factors that contribute to this gap in care include: the need to translate adolescent blood pressure (BP) measures into blood pressure percentiles on the basis of age, gender, and height, lack of familiarity with National High Blood Pressure Education Program (NHBPEP) clinical guidelines, and competing demands at clinical encounters.

Electronic health record (EHR)-based clinical decision support (CDS) can be used to address these barriers and support better care of elevated blood pressure (BP) and Hypertension (HT) in adolescents. In this project, the investigators integrate EHR-extracted data with sophisticated Web-based CDS algorithms to provide patient-specific point-of-care clinical recommendations, in accordance with NHBPEP guidelines. To evaluate the impact of this innovation on quality and cost of care, the investigators randomize 18 clinics with their 130 pediatric care providers (PCP) and their estimated 17,000 adolescent patients to receive or not receive this EHR-based CDS intervention. The investigators hypothesize that the intervention will improve recognition and early management of elevated BP and that short-term increases in outpatient care costs will be offset by longer-term clinical benefits, estimated using established econometric models.

This innovative project (a) addresses the under-recognized high-risk patient population of adolescents, (b) integrates EHR and Web-based CDS technology to provide sophisticated patient-specific point-of-care CDS, (c) develops and implements novel and intuitive visual interfaces to communicate CDS recommendations to PCPs, and (d) provides both clinical and cost outcome data useful to clinicians and policymakers. If the EHR-based CDS intervention improves adherence to NHBPEP recommendations, it will provide a much-needed tool to combat the burgeoning problem of rising cardiovascular risk factors in children and adolescents. Further, regardless of outcome, the technology that is developed and tested will provide many useful insights to advance the science of EHR-based CDS. This will, in turn, help translate the massive public and private investments in EHR technology into improved adolescent health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents age 10-17
* Pediatric and Family Medicine Providers

Exclusion Criteria:

* Pregnant adolescents
* Within 12 weeks post partum

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31579 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04-16 (Actual); Study Completion 2017-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elyse O Kharbanda, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Medical Group, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] National High Blood Pressure Education Program Working Group on High Blood Pressure in Children and Adolescents. The fourth report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. Pediatrics. 2004 Aug;114(2 Suppl 4th Report):555-76. No abstract available. PMID 15286277
- [Derived] Kharbanda EO, Asche SE, Sinaiko AR, Ekstrom HL, Nordin JD, Sherwood NE, Fontaine PL, Dehmer SP, Appana D, O'Connor P. Clinical Decision Support for Recognition and Management of Hypertension: A Randomized Trial. Pediatrics. 2018 Feb;141(2):e20172954. doi: 10.1542/peds.2017-2954. PMID 29371241

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary care providers (physicians, physician assistants,nurse practitioners) as of April 2014 were eligible. Providers received a letter inviting them to complete surveys (pre and post intervention). Completing surveys was considered implied consent. Patient consent was waived as no direct contact between patients and study team occurred.
Pre-assignment Details: 31,579 patients 10-17 years of age with >=1 BP measurement were assessed for eligibility for the primary analysis. After excluding for non-incident hypertension, and restricting to patients with BPs at >=3 visits with BP >=95th percentile who meet case definitions for new onset hypertension, the analytic denominator equals 522.
Groups:
- Clincal Decision Support (CDS): The Clinical Decision Support (CDS) tool will be activated when a BP is entered in the vital sign section of the electronic health record (EHR). Data is exchanged between the EHR and the CDS that runs the data through algorithms and returns a response with appropriate action to the EHR. The CDS tool, includes six key features: (i) prompts regarding the need for height data to classify the BP by percentile (ii) prompts to repeat any BP that is ≥90% or ≥120/80 mm Hg (iii) classification of BPs by percentile, including classification of those in pre-hypertension, stage 1 hypertension and stage 2 hypertension range (iv) review of previous hypertension diagnoses and BPs in order to classify elevated BPs as incident (first or second elevated BP) or persistent (third or greater elevated BP) (v) tailored CDS based on hypertension category and previous diagnoses (vi) graphical representation of current and historical BP data by age and BP percentile.
Period: Overall Study
Arm/Group | Clincal Decision Support (CDS) | Control
Started | 17037 | 14542
Completed | 296 | 226
Not Completed | 16741 | 14316

BASELINE CHARACTERISTICS:
Groups:
- Clincal Decision Support (CDS): The Clinical Decision Support (CDS) tool will be activated when a BP is entered in the vital sign section of the EHR. Data is exchanged between the EHR and the CDS that runs the data through algorithms and returns a response with appropriate action to the EHR. The CDS tool, called Peds & TeenBP, includes six key features: (i) prompts regarding the need for height data to classify the BP by percentile (ii) prompts to repeat any BP that is ≥90% or ≥120/80 mm Hg (iii) classification of BPs by percentile, including classification of those in pre-HT, stage 1 HT and stage 2 HT range (iv) review of previous HT diagnoses and BPs in order to classify elevated BPs as incident (first or second elevated BP) or persistent (third or greater elevated BP) (v) tailored CDS based on HT category and previous diagnoses (vi) graphical representation of current and historical BP data by age and BP percentile.
- Total: Total of all reporting groups
Arm/Group | Clincal Decision Support (CDS) | Control | Total
Number analyzed (Participants) | 296 | 226 | 522
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.5 (2.1) | 14.4 (2.0) | 14.5 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 125 | 296
  Male | 125 | 101 | 226
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 14 | 42
  Not Hispanic or Latino | 268 | 212 | 480
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 8 | 17
  Asian | 25 | 25 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 53 | 45 | 98
  White | 195 | 131 | 326
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 16 | 30
Region of Enrollment [Number; unit: participants]
  United States | 296 | 226 | 522
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  Body Mass Index <85th | 104 | 68 | 172
  Body Mass Index 85-<=95th | 67 | 51 | 118
  Body Mass Index >=95th | 125 | 107 | 232

OUTCOME MEASURES:

1. Primary Outcome: Participants With Clinical Recognition of Hypertension
Description: Clinical recognition of hypertension as determined by one or more of the following; 1) hypertension or elevated BP as discharge diagnosis, 2) hypertension or elevated BP in the clinical note, 3) hypertension or elevated BP in discharge instructions, 4) hypertension or elevated BP added to the problem list.
Time Frame: 6 months
Population: The sample was restricted to patients with blood pressures at >=3 visits with blood pressure >=95th percentile, who were then passively monitored for study endpoints. Patients with a previous hypertension diagnosis were excluded.
Measure: Count of Participants; unit: Participants
Groups:
- Clinical Decision Support (CDS): The Clinical Decision Support (CDS) tool will be activated when a BP is entered in the vital sign section of the EHR. Data is exchanged between the EHR and the CDS that runs the data through algorithms and returns a response with appropriate action to the EHR. The CDS tool, called Peds & TeenBP, includes six key features: (i) prompts regarding the need for height data to classify the BP by percentile (ii) prompts to repeat any BP that is ≥90% or ≥120/80 mm Hg (iii) classification of BPs by percentile, including classification of those in pre-HT, stage 1 HT and stage 2 HT range (iv) review of previous HT diagnoses and BPs in order to classify elevated BPs as incident (first or second elevated BP) or persistent (third or greater elevated BP) (v) tailored CDS based on HT category and previous diagnoses (vi) graphical representation of current and historical BP data by age and BP percentile.
Arm/Group | Clinical Decision Support (CDS) | Control
Number analyzed (Participants) | 296 | 226
Participants | 160 | 51
Statistical Analysis 1: Comparison: Clinical Decision Support (CDS) vs Control; Test type: Superiority; p < .001, Mixed Models Analysis; Odds Ratio (OR) = 4.51

2. Primary Outcome: Participants With Appropriate Workup for Secondary Causes of Hypertension
Description: Appropriate workup for those with incident hypertension included an initiated workup for secondary causes of hypertension or end organ damage, defined as referral to cardiology, nephrology, or endocrinology, and/or orders for echocardiogram, ECG, or renal ultrasound.
Time Frame: 6 months
Population: The sample was restricted to patients with BPs at >=3 visits with BP >=95th percentile, who were then passively monitored for study endpoints. Patients with a previous HT diagnosis were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Clincal Decision Support (CDS) | Control
Number analyzed (Participants) | 296 | 226
Participants | 29 | 10
Statistical Analysis 1: Comparison: Clincal Decision Support (CDS) vs Control; Test type: Superiority; p = .046, Mixed Models Analysis; Odds Ratio (OR) = 2.36

3. Primary Outcome: Participants With Appropriate Lifestyle Referral
Description: Appropriate lifestyle referral is defined as referral to dietitian, weight loss, or exercise program within 6 months of meeting criteria for incident hypertension.
Time Frame: 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Clincal Decision Support (CDS) | Control
Number analyzed (Participants) | 296 | 226
Participants | 55 | 10
Statistical Analysis 1: Comparison: Clincal Decision Support (CDS) vs Control; Test type: Superiority; p = .001, Mixed Models Analysis; Odds Ratio (OR) = 5.13

ADVERSE EVENTS:
Time Frame: Safety events were passively monitored every 6 months during the 2 year intervention period. Patients were monitored for events occurring within 3 months of meeting hypertension criteria.
Description: We conducted passive safety surveillance for patients in control and intervention sites using routinely collected electronic health record data to monitor for potential safety events. Neurological complications were not identified but include increased intracranial pressure, hypertensive encephalopathy, or cerebral edema at any point during the intervention period. Since no cases were identified, they are pooled here for the sake of simplicity.
Arm/Group | Clincal Decision Support (CDS) | Control
Serious Adverse Events (participants affected / at risk) | 2/296 | 1/226
Other Adverse Events (participants affected / at risk) | 32/296 | 15/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clincal Decision Support (CDS) (N=296) | Control (N=226)
Very high blood pressure (Vascular disorders) | 2 | 1 — Blood pressure greater than 160/100 at any point in the intervention period.
Stroke/transient ischemic attack (TIA) (Vascular disorders) | 0 | 0 — Stroke or TIA occurring in any point during the intervention period.
Acute renal failure (Renal and urinary disorders) | 0 | 0 — Acute renal failure at any point during the intervention period.
Neurological complications (Nervous system disorders) | 0 | 0 — Neurologic complications were pooled as none were identified. They include increased intracranial pressure, hypertensive encephalopathy, or cerebral edema at any point during the intervention period.
Hypertensive retinopathy (Eye disorders) | 0 | 0 — Hypertensive retinopathy at any point during the intervention period.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clincal Decision Support (CDS) (N=296) | Control (N=226)
Elevated serum creatinine (Renal and urinary disorders) | 3 | 3
Echocardiogram conducted (Surgical and medical procedures) | 7 | 1
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0
Renal ultrasound conducted (Surgical and medical procedures) | 8 | 2
Abnormality on renal ultrasound (Renal and urinary disorders) | 0 | 0
New medication for hypertension (Vascular disorders) | 3 | 1
Hospitalization for any cause (General disorders) | 11 | 8

LIMITATIONS AND CAVEATS:
Because this study was conducted at a single medical group, generalizability of results to other care delivery systems or patient populations is uncertain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No